CLINICAL TRIAL: NCT00936611
Title: Phase II Trial of LBH589 (Panobinostat) in Relapsed or Relapsed and Refractory Waldenstrom's Macroglobulinemia
Brief Title: LBH589 in Relapsed or Relapsed and Refractory Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-071; CLBH589CUS56T (Other: Novartis)
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: LBH589; WM; panobinostat; relapsed; waldenstrom; macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Recurrence | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LBH589 (Experimental): 30 mg three days a week (Mondays, Wednesdays and Fridays).
  1 cycle was 28 days
  Dose modifications for attributable toxicities allowed for reduction to:
  * 25 mg, 20 mg three times a week every week
  * Or 20 mg three times a week every other week. No dose re-escalation was allowed.
    * The protocol was amended on 6/15/2010 because of concerns of toxicity to allow a starting dose of 25 mg; 12/36 (33%) patients were enrolled on the 25 mg dose.
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589
  Other Names: panobinostat

SUMMARY:
The purpose of this research study is to assess the overall response rate of LBH589 in patients with relapsed or refractory Waldenstrom's Macroglobulinemia. LBH589 is a newly discovered compound that has killed Waldenstrom cells in laboratory studies, however, it is not known if LBH589 will show the same activity in people with Waldenstrom's Macroglobulinemia. This drug has been used in research for the treatment of other types of cancer, such as multiple myeloma.

DETAILED DESCRIPTION:
This phase II study is designed to assess the toxicity profile and the proportion of overall response in patients with relapsed or refractory WM. This will study the effect of single agent LBH589 on response in these patients. Efficacy measures will include both objective clinical measurements and investigator-reported outcomes. Response and time to event analyses will follow the criteria set forth in the International Waldenstrom consortium recommendations. Prior to the start of the study, investigators will assess disease and perform a CT scan of the chest, abdomen and pelvis.

Response will be assessed after 2 cycles. If patients have stable disease or response, then they will continue on therapy until progression or unacceptable toxicity, being assessed every cycle until the sixth cycle and then every 3 months. Patients who show progression after 2 cycles will come off therapy and undergo event monitoring every 3 months. All responses will be assessed by M-protein quantification and immunofixation from serum and IgM monoclonal protein level. In addition, BM biopsies will be done at baseline, at the end of cycle 6 and at the end of all therapy. The protocol was amended because of concerns of toxicity to allow a starting dose of 25 mg; 12/36 (33%) patients were enrolled on the 25 mg dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older
* Must have received prior therapy for their WM, any number of prior therapies is allowed
* Must have symptomatic relapsed or refractory WM
* Measurable monoclonal IgM protein in the blood and presence of lymphoplasmacytic cells in the bone marrow during any previous bone marrow
* Laboratory values as described in the protocol
* Clinically euthyroid
* ECOG Performance Status of 2 or less

Exclusion Criteria:

* Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment
* Peripheral neuropathy CTCAE grade 2 or higher
* Impaired cardiac function or clinically significant cardiac diseases
* Impairment of GI function or GI disease that may significantly alter the absorption of LBH589
* Diarrhea > CTCAE grade 1
* Other concurrent severe and/or uncontrolled medical conditions including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
* Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Patients who have received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is longer) and who have not recovered from side effects of those therapies
* Patients who have received chemotherapy or rituximab within 3 weeks or less; or radiation therapy to > 30% of marrow-bearing bone within 2 weeks or less prior to starting study treatment; or who have not yet recovered from side effects of such therapies
* Patients who have received corticosteroids 2 weeks or less prior to registration. Patients may be receiving chronic corticosteroids if they are being given for disorders other than than Waldenstrom's Macroglobulinemia
* Patients with active bleeding tendency or receiving any treatment with therapeutic doses of sodium warfarin or coumadin derivatives. Low doses of Coumadin to maintain line patency is allowed
* Patients who have undergone major surgery 4 weeks or less prior to starting study drug or who have not recovered from side effects of such therapy
* Women who are pregnant or breast feeding or women of childbearing potential not using an effective method of birth control
* Male patients whose sexual partners are women of childbearing potential not using effective methods of birth control
* Patients with prior malignancy within the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients with a significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Ghobrial IM, Campigotto F, Murphy TJ, Boswell EN, Banwait R, Azab F, Chuma S, Kunsman J, Donovan A, Masood F, Warren D, Rodig S, Anderson KC, Richardson PG, Weller E, Matous J. Results of a phase 2 trial of the single-agent histone deacetylase inhibitor panobinostat in patients with relapsed/refractory Waldenstrom macroglobulinemia. Blood. 2013 Feb 21;121(8):1296-303. doi: 10.1182/blood-2012-06-439307. Epub 2013 Jan 3. PMID 23287861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2009 to March 2011
Groups:
- LBH589: 30 mg three days a week (Mondays, Wednesdays and Fridays).
  1 cycle was 28 days
  Dose modifications for attributable toxicities allowed for reduction to:
  * 25 mg, 20 mg three times a week every week
  * Or 20 mg three times a week every other week. No dose re-escalation was allowed.
    * The protocol was amended on 6/15/2010 because of concerns of toxicity to allow a starting dose of 25 mg; 12/36 (33%) patients were enrolled on the 25 mg dose.
  LBH589
Period: Overall Study
Arm/Group | LBH589
Started | 39
Treated (3 patients deemed ineligible) | 36
Starting Dose Reduction: 30 mg to 25 mg (Protocol Amendment 6/15/2010. Study drug starting dose reduced.) | 12
Completed (Since treatment was not of fixed duration, all participants were considered as 'Not Completed' and reason off-treatment is provided.) | 0
Not Completed | 39
Not completed — Progressive Disease | 3
Not completed — New Systemic Therapy | 22
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Still on Follow-up | 1
Not completed — Still on Active Therapy | 7
Not completed — Ineligible for Study Drug | 3

BASELINE CHARACTERISTICS:
Arm/Group | LBH589
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 61.6 [47 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 1
Median IgM [Median (Full Range); unit: mg/dL] | 3240 [804 to 10300]
Median M Spike [Median (Full Range); unit: gm/dL] | 2.06 [0.63 to 5.1]
Median Platelets [Median (Full Range); unit: platelets x 10^3 / mL] | 242 [74 to 388]
Median Hemoglobin [Median (Full Range); unit: gm/dL] | 10.7 [8.2 to 14.5]
Median Beta 2 Microglobulin [Median (Full Range); unit: mg/dL] | 3.3 [1.4 to 7.4]
Percentage of Bone Marrow Involvement [Median (Full Range); unit: percentage of marrow] | 70 [5 to 100]
Lymph Nodes and Hepatocyte Selection Medium Assessment by CT Scan Evidence of Disease [Count of Participants; unit: Participants]
  Present | 29
  Absent | 7
International Prognostic Scoring System for Waldenstrom Macroglobulinemia [Count of Participants; unit: Participants] — Measure Description: Low is defined as 1 or dewer of the following:
  Hemoglobin (HB) <=11.5 g/dL Platelet (PT) <=100 x 10^9 / L Beta 2 Microglubin (B2M) > 3 mg/L Immunoglobulin M (IgM) > 7 g/dL
  Intermediate is defined as over 65 years old or two of the following:
  HB <=11.5 g/dL PT <=100 x 10^9 / L B2M > 3 mg/L IgM> 7 g/dL
  High is defined as more than 2 of the following:
  Over 65 years old HB <=11.5 g/dL PT <=100 x 10^9 / L B2M > 3 mg/L IgM> 7 g/dL
  Participants
    High | 7
    Intermediate | 14
    Low | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate is percentage of participants with complete (CR), very good partial (VGPR), partial (PR), or minimal response (MR) as best response during treatment.
  CR
  * Disappearance of monoclonal protein by immunofixation
  * No histologic evidence of bone marrow involvement
  * Resolution of any adenopathy/organomegaly (confirmed by CT scan), or signs or symptoms attributable to WM.
  * Second immunofixation required for confirmation.
  VGPR
  -At least 90% reduction of serum monoclonal IgM concentration on protein electrophoresis.
  PR
  * At least 50% reduction of serum monoclonal IgM concentration on protein electrophoresis and at least 50% decrease in adenopathy/organomegaly on physical examination or on CT scan.
  * No new symptoms or signs of active disease.
  MR
  * At least 25% but less than 50% reduction of serum monoclonal IgM by protein electrophoresis.
  * No new symptoms or signs of active disease.
Time Frame: Assessed after 2nd cycle and then every subsequent cycle for 6 cycles. The median number of completed cycles of therapy was 5 (0- 32). As such observed up to ~32 months.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | LBH589
Number analyzed (Participants) | 36
percentage of participants | 47 [33 to 62]

2. Secondary Outcome: Median Progression Free Survival
Description: Progression free survival (PFS) is defined as the time from start of treatment to disease progression or death from any cause as estimated by Kaplan Meier methods. Patients who have not progressed and are alive are censored at the date the patient is known to be progression-free.
Time Frame: Assessed after 2nd cycle and then every subsequent cycle for 6 cycles and then every 3 months. If taken off treatment at cycle 2 for disease progression, assessed every 3 months. The median (range) follow up from treatment start is 7.7 month (0.9 - 29.7).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LBH589
Number analyzed (Participants) | 36
months | 6.6 [5.5 to 14.8]

3. Secondary Outcome: Median Time to Progression
Description: Time to progression (TTP) is defined as the time from start of treatment to progression. Patients who have not progressed are censored at the date the patient is last known to be progression free.
Time Frame: as for outcome 2
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LBH589
Number analyzed (Participants) | 36
months | 6.6 [5.5 to 14.8]

4. Secondary Outcome: Median Duration of Response
Description: Duration of response DR is defined as the time from the date of first response after treatment to the date of disease progression Patients who have died for any cause or are alive without progression are censored at the date the patient is last know to be progression-free.
  Duration of response DR is defined as the time from the date of first response after treatment to the date of disease progression or death for any cause. Patients who are alive without progression are censored at the date the patient is last know to be progression-free.
Time Frame: as for outcome 2
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LBH589
Number analyzed (Participants) | 36
months | 6.9 [3.1 to 18.9]

5. Secondary Outcome: Number of Participants With Grade 3 and 4 Treatment-Related Thrombocytopenia
Description: Grade 3 thrombocytopenia is defined as having 25,000-50,000 /uL platelets
  Grade 4 thrombocytopenia is defined as having < 25,000 /uL platelets
Time Frame: Assessed after 2nd cycle, every subsequent cycle for 6 cycles and then every 3 months. Once off-treatment, adverse events will be assessed for 30 days. The median (range) number of completed cycles of therapy was 5 (0- 32). Therefore, up to ~33 months.
Measure: Number; unit: participants
Arm/Group | LBH589
Number analyzed (Participants) | 36
participants | 24

6. Secondary Outcome: Acetylated Histone H3 and Overall Response Association
Description: Acetylated-histone-H3 levels were obtained through bone marrow biopsies and measured using established methods. This analysis aimed to analyze the association between overall response and percent change of acetylated histone h3 in samples using a paired t-test.
Time Frame: Bone marrow biopsies were obtained at the start of treatment (baseline) and after the 6th cycle.
Population: Only three complete sample (baseline and post-therapy) were ascertained. The difference in percentage of acetylated histone h3 were not large enough to conduct the correlative analysis.
Arm/Group | LBH589
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Assessed after 2nd cycle, every subsequent cycle for 6 cycles and then every 3 months. Once off-treatment, adverse events will be assessed for 30 days. The median (range) number of completed cycles of therapy was 5 (0- 32). Therefore, up to ~33 months.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | LBH589
All-Cause Mortality (participants affected / at risk) | 28/39
Serious Adverse Events (participants affected / at risk) | 29/39
Other Adverse Events (participants affected / at risk) | 36/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LBH589 (N=39)
Hemoglobin (Blood and lymphatic system disorders) | 10
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Lower GI, hemorrhage NOS (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 5
Infection w/ unk ANC lung (Infections and infestations) | 1
Leukocytes (Investigations) | 7
Neutrophils (Investigations) | 13
Platelets (Investigations) | 23
Bilirubin (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 2
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LBH589 (N=39)
Infection w/ gr3-4 neut, upper airway (Infections and infestations) | 1
Infection Gr0-2 neut, dental-tooth (Infections and infestations) | 1
Infection Gr0-2 neut, sinus (Infections and infestations) | 2
Infection Gr0-2 neut, upper airway (Infections and infestations) | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1
Infection w/ unk ANC middle ear (Infections and infestations) | 1
Intra-op injury Other (Specify) (Injury, poisoning and procedural complications) | 1
Hemoglobin (Blood and lymphatic system disorders) | 14
Lymph node, pain (Blood and lymphatic system disorders) | 2
Palpitations (Cardiac disorders) | 4
Sinus tachycardia (Cardiac disorders) | 2
Cardiac-other (Cardiac disorders) | 1
Hearing w/w-o audiogr in monitor prg (Ear and labyrinth disorders) | 1
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 1
Middle ear, pain (Ear and labyrinth disorders) | 3
Dry eye syndrome (Eye disorders) | 1
Vision-blurred (Eye disorders) | 3
Tearing (Eye disorders) | 1
Ocular-other (Eye disorders) | 1
Eye, pain (Eye disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Periodontal disease (Gastrointestinal disorders) | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 21
Dry mouth (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 3
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 6
GI-other (Gastrointestinal disorders) | 2
Lower GI, hemorrhage NOS (Gastrointestinal disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 7
Anus, pain (Gastrointestinal disorders) | 1
Stomach, pain (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 28
Fever w/o neutropenia (General disorders) | 4
Rigors/chills (General disorders) | 2
Edema limb (General disorders) | 8
Chest/thoracic pain NOS (General disorders) | 4
Flu-like syndrome (General disorders) | 1
Allergy-other (Immune system disorders) | 1
Infection w/ gr3-4 neut, skin (Infections and infestations) | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 1
Infection Gr0-2 neut, sinus (Infections and infestations) | 1
Infection-other (Infections and infestations) | 3
Bruising (Injury, poisoning and procedural complications) | 3
Leukocytes (Investigations) | 18
Neutrophils (Investigations) | 21
Platelets (Investigations) | 16
Weight loss (Investigations) | 8
Bilirubin (Investigations) | 1
Creatinine (Investigations) | 5
Pancreatic glucose intolerance (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 16
Dehydration (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 2
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 5
Joint, pain (Musculoskeletal and connective tissue disorders) | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 3
Neck, pain (Musculoskeletal and connective tissue disorders) | 3
Taste disturbance (Nervous system disorders) | 11
Cognitive disturbance (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 7
Neuropathy-sensory (Nervous system disorders) | 5
Tremor (Nervous system disorders) | 2
Neurologic-other (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 6
Sinus, pain (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Urethra, pain (Renal and urinary disorders) | 1
Obstruction-ureteral (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 5
Sweating (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 6
Nail changes (Skin and subcutaneous tissue disorders) | 4
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Skin-other (Skin and subcutaneous tissue disorders) | 2
Petechiae (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT00936611/Prot_SAP_000.pdf